CLINICAL TRIAL: NCT05103735
Title: Propofol-remifentanil Versus Dexmedetomidine in Awake Craniotomy: an Intraoperative Neurophysiological Evaluation
Brief Title: Propofol-remifentanyl Versus Dexmedetomidine in Awake Craniotomy: Impact on Electroclinical Seizure Activity
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Cristian Deana, Principal Investigator, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: CRANIO-UDINE
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Craniotomy; Seizures; Dexmedetomidine; Propofol; Remifentanil; Cerebral Tumor; Neurophysiology
MeSH Terms: conditions — Seizures | interventions — Propofol; Remifentanil; Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PROPOFOL-REMIFENTANYL: Awake craniotomy under propofol-remifentanil sedation. Propofol and remifentanyl was administered through continuous intravenous infusion, starting 30 minutes prior to surgery. The end of the infusion was at the end of the surgical procedure.
  Propofol dosage: 0.2-2 mk/kg/h Remifentanyl dosage: 0.01-0.1 mcg/kg/min
  Interventions: Drug: Propofol
- DEXMEDETOMIDINE: Awake craniotomy under dexmedetomidine sedation. Dexmedetomidine was administered through continuous intravenous infusion, starting 30 minutes prior to surgery. The end of the infusion was at the end of the surgical procedure.
  Dexmedetomidine dosage: 0.2-1 mcg/kg/h In this group, remifentanyl administration was allowed.

INTERVENTIONS:
Drug: Propofol — awake neurosurgery under propofol-remifentanil sedation
  Other Names: Remifentanil; Dexmedetomidine
  Groups: PROPOFOL-REMIFENTANYL

SUMMARY:
Awake craniotomy require a cooperative patient during resection neurosurgery phase. Anesthesiologist should guarantee analgesia, sedation, nausea and vomiting prevention, while maintaining normal vital parameters.

Neurosurgeon could be help by Intraoperative electrocorticography to maximise lesion resection and avoiding neurologic sequelae. Propofol and remifentanyl have been largely used. Dexmedetomidine represents an alternative. However little is known about the role of dexmedetomidine on Intraoperative electrocorticography.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS UNDERGOING AWAKE CRANIOTOMY FOR TUMOR RESECTION (EXCLUDED E.G. SURGERY OF EPILEPSIA)
* INTRAOPERATIVE MONITORING (IOM) WITH ELECTROCORTICOGRAPHY
* AWAKE-AWAKE-AWAKE TECHNIQUE

Exclusion Criteria:

* AGE <18 YEARS OLD
* NON AWAKE-AWAKE-AWAKE TECHNIQUE
* ABSENCE OF IOM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL PATIENTS UNDERGOING AWAKE CRANIOTOMY FOR TUMOR RESECTION SURGERY
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
SEIZURE ACTIVITY | DURING TUMOR RESECTION PHASE OF THE AWAKE CRANIOTOMY
  INCIDENCE OF ELECTRO-CLINICAL SEIZURE ACTIVITY IN THE TWO GROUPS DURING RESECTIVE PHASE OF AWAKE CRANIOTOMY EVALUATED WITH ELECTROCORTICOGRAPHY.

CONTACTS AND LOCATIONS:
Locations (1):
- Cristian Deana, Udine, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Deana C, Pez S, Ius T, Furlan D, Nilo A, Isola M, De Martino M, Mauro S, Verriello L, Lettieri C, Tomasino B, Valente M, Skrap M, Vetrugno L, Pauletto G. Effect of Dexmedetomidine versus Propofol on Intraoperative Seizure Onset During Awake Craniotomy: A Retrospective Study. World Neurosurg. 2023 Apr;172:e428-e437. doi: 10.1016/j.wneu.2023.01.046. Epub 2023 Jan 20. PMID 36682527